CLINICAL TRIAL: NCT01713465
Title: An Innovative Informatics Platform to Deliver a Multidimensional Intervention to Prevent and Manage Metabolic Syndrome
Brief Title: Use of Computers to Prevent Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Public Health (Other)
Responsible Party: Principal Investigator, Ashish Joshi, Assistant Professor, Asian Institute of Public Health
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: GIA22012
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Metabolic Syndrome
Keywords: Diabetes; Hypertension; Hypercholesterolemia; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Hypertension; Hypercholesterolemia; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 CBMP (Experimental): CBMP: Computer based Metabolic syndrome program
  Interventions: Other: Computer based Metabolic Syndrome educational program

INTERVENTIONS:
Other: Computer based Metabolic Syndrome educational program — Individuals in the intervention group will receive metabolic syndrome related education using a touch screen interactive and bilingual multimedia enabled educational program
  Other Names: CBMP

SUMMARY:
The objective of the proposed study is to design and evaluate a touch screen computer based multi-factorial intervention to educate individuals at risk of Metabolic syndrome in diverse Indian settings including urban, rural and slum in the State of Bhubaneshwar. The study objective is to improve metabolic syndrome related knowledge, attitude and practices among individuals using the proposed interactive, bilingual computer based educational program.

DETAILED DESCRIPTION:
The rising prevalence of overweight and obesity has a direct correlation with increasing prevalence of hypertension, dyslipidemia, type2 diabetes mellitus (T2DM), Metabolic Syndrome (MetS), and Cardiovascular diseases (CVD). Most of the previous studies in India have been cross sectional nature and have looked at prevalence of Metabolic Syndrome (MetS. Despite the clinical and public health importance of this phenomenon, not enough work has been carried out so far to study and remedy this situation. A computer based interactive and bilingual system is proposed to improve Metabolic syndrome related knowledge, attitudes and practices among individuals living in urban, rural and slum settings of Bhubaneswar, India. We propose to enroll 750 individuals and the eligible study participants will be randomly assigned to either the intervention (computer based MetS Program CBMP) or control (Printed Educational Material, PEM) groups. The study participants will be followed at days 30, 60 and 90 days following the baseline visit. The primary outcomes include change in knowledge, attitudes and practices and secondary outcomes include improvement in quality of life and increase satisfaction to medical care.

ELIGIBILITY:
Inclusion Criteria:

* adults age 30 years and above, agreeing to participate in the study available for follow-up interview.

Exclusion Criteria:

* mental and physical challenge that makes it difficult to use the touch based computer program nonavailability for telephone follow-up involvement in other clinical trials or protocols related to Metabolic Syndrome.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-01 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of participants with increase in Knowledge, Attitude and Practice scores | 3 months
Frequency of participants with increase in treatment adherence scores | 3 months

SECONDARY OUTCOMES:
Frequency of participants with increase in Satisfaction to Medical Care | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Joshi, MD,PhD, MPH, Principal Investigator — UNMC
Locations (1):
- Center for Public Health informatics, AIPH, Bhubaneshwar, Odisha, India

REFERENCES:
- [Background] Finkelstein J, Joshi A, Hise MK. Association of physical activity and renal function in subjects with and without metabolic syndrome: a review of the Third National Health and Nutrition Examination Survey (NHANES III). Am J Kidney Dis. 2006 Sep;48(3):372-82. doi: 10.1053/j.ajkd.2006.05.013. PMID 16931210
- [Derived] Joshi A, Mehta S, Talati K, Grover A. Protocol for an experimental study design to evaluate computer-enabled intervention to prevent and manage metabolic syndrome. BMJ Open. 2013 Mar 1;3(3):e002163. doi: 10.1136/bmjopen-2012-002163. PMID 23454666